CLINICAL TRIAL: NCT03278574
Title: Mitral Valve Repair Using Flexible Bands Versus Complete Rings in Patients With Degenerative Mitral Valve Disease: a Prospective, Randomized Study
Brief Title: Flexible Band vs Rigid Ring for Degenerative Mitral Valve Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25041214
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible band (Experimental): Mitral valve repair with flexible posterior annuloplasty band
  Interventions: Procedure: Mitral valve repair; Device: Ring annuloplasty with posterior band
- Complete ring (Active Comparator): Mitral valve repair with complete rigid ring
  Interventions: Procedure: Mitral valve repair; Device: Ring annuloplasty with complete ring

INTERVENTIONS:
Procedure: Mitral valve repair — Mitral valve repair with standard technique: resection of prolapsed leaflet and/or artificial neochordae implantation
Device: Ring annuloplasty with posterior band — Mitral valve annuloplasty using Cardiamed (Penza, Russia) flexible posterior annuloplasty band
  Arms: Flexible band
Device: Ring annuloplasty with complete ring — Mitral valve annuloplasty using Cardiamed (Penza, Russia) complete semirigid ring
  Arms: Complete ring

SUMMARY:
The study evaluates the results of mitral valve repair with flexible band in comparison with rigid ring in patients undergoing mitral valve repair for degenerative mitral valve disease

DETAILED DESCRIPTION:
Currently, mitral ring selection is based on a surgeon's preference rather than evidence. Semirigid rings combine flexibility and stability; however, their clinical benefit has not been completely clarified. The present study aimed to compare the outcomes of mitral valve repair with a flexible posterior annuloplasty band versus complete semirigid ring in patients with degenerative mitral valve disease.

ELIGIBILITY:
Inclusion Criteria:

* severe primary mitral regurgitation due to degenerative mitral valve disease

Exclusion Criteria:

* previous open cardiac surgery,
* indication for concomitant aortic valve replacement,
* left ventricle impairment (ejection fraction < 40%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2014-09-29 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
Freedom from significant mitral regurgitation | 12 months
  Significant mitral regurgitation is defined as moderate and severe mitral regurgitation. The severity of MR was evaluated and defined in accordance with the European Association of Echocardiography recommendations for the assessment of valvular regurgitation

SECONDARY OUTCOMES:
Survival | 12 months, 24 months
  Continued existence at follow up
Freedom from reoperations | 12 months, 24 months
  Freedom from redo mitral valve surgery during follow up
Freedom from severe MR recurrence | 12 months
  The severity of MR was evaluated and defined in accordance with the European Association of Echocardiography recommendations for the assessment of valvular regurgitation

IPD SHARING:
Plan to Share IPD: No
individual participant data is unavailable for security reason

REFERENCES:
- [Derived] Bogachev-Prokophiev AV, Afanasyev AV, Zheleznev SI, Nazarov VM, Sharifulin RM, Karaskov AM. Mid-term results of mitral valve repair using flexible bands versus complete rings in patients with degenerative mitral valve disease: a prospective, randomized study. J Cardiothorac Surg. 2017 Dec 13;12(1):113. doi: 10.1186/s13019-017-0679-0. PMID 29237465